CLINICAL TRIAL: NCT04111250
Title: Crestal Versus Lateral Sinus Lift: One-year Results From a Within-patient Randomised Controlled Trial
Brief Title: Crestal vs Lateral Sinus Lift Augmentation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital San Pietro Fatebenefratelli (Other)
Responsible Party: Principal Investigator, Marco Tallarico, Lecturer, Hospital San Pietro Fatebenefratelli
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: iRaise_RCT
Record Dates: First submitted 2019-06-16; First posted 2019-10-01 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Edentulous Alveolar Ridge; Bone Atrophy, Alveolar
Keywords: Dental implants; Maxillary sinus augmentation; Crestal approach
MeSH Terms: conditions — Alveolar Bone Loss | interventions — Sinus Floor Augmentation

STUDY DESIGN:
Intervention Model Description: Split mouth design
Who Masked: Outcomes Assessor
Masking Description: Where possible, outcomes assessor was blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Crestal sinus lift using iRasie implant (Experimental): Device: iRaise Sinus Lift implant (Maxillent, Herzliya, Israel). Procedure: crestal sinus lift augmentation.
  We tested crestal versus lateral approach to the sinus. Crestal approach is made by a novel device (iRaise, implant system). Lateral approach is made conventionally with gold standard procedure (lateral approach).
  The iRaise Sinus Lift implant is made of Titanium-6 Aluminum-4 Vanadium alloy, have a surface treated with grit blasting using an apatitic calcium phosphate media, followed by acid etching, and have an internal hexagon connection. Implants have an internal l-shape channel to allow saline and graft passage.
  This implants system is made to perform crestal sinus lift procedure at the same time of the implant placement using the same device. After implant site preparation and initial implant placement, the hydraulic system is connected to the implant to allow the injection of saline and then graft the material. Then, the implant, is inserted for its full length.
  Interventions: Procedure: Maxillary sinus augmentation
- Lateral sinus lift (Active Comparator): Conventional procedure.
  Lateral approach to the sinus was made following the conventional procedure.
  A window on the lateral wall of the sinus is performed according to a conventional surgical lateral approach to the sinus cavity. Graft materials is filled inside the sinus cavity. Finally, iSure implants [Maxillent] are placed, and flap is sutured.
  Interventions: Procedure: Maxillary sinus augmentation

INTERVENTIONS:
Procedure: Maxillary sinus augmentation — Raise the sinus membrane to graft bone substitute to augment the sinus cavity allowing implants placement.
  Other Names: Sinus lift

SUMMARY:
The aim of this randomised controlled trial (RCT) of split-mouth design was to compare patient preference and effectiveness of two different techniques for lifting the maxillary sinus: the crestal approach versus the lateral window approach.

DETAILED DESCRIPTION:
Each patient having bilateral edentulism in posterior maxillae was randomised to receive one partial fixed prosthesis supported by one to three implants placed either with a crestal or with lateral window sinus lift procedure.

Eligibility criteria for participants

Only healed implant sites were considered (at least 3 months after tooth extraction). The vertical bone height at the implant sites to be included had to be between 2 to 6 mm and bone thickness at least 6 mm as measured on cone-bean computed tomography (CBCT) scans.

Patients were not admitted in the study if any of the following exclusion criteria was present:

general contraindications to implant surgery subjected to irradiation in the head and neck area immunosuppressed or immunocompromised treated or under treatment with intravenous amino-bisphosphonates poor oral hygiene and motivation untreated periodontal disease uncontrolled diabetes pregnant or lactating substance abusers psychiatric problems unrealistic expectations lack of opposite occluding dentition/prosthesis in the area intended for implant placement acute or chronic infection/inflammation in the area intended for sinus augmentation/implant placement referred only for implant placement who cannot be rehabilitated and followed at the treatment centre unable to attend a 5-year post-loading follow-up. Smokers were included and patients were categorised into three groups according to what declare: i) non-smokers; ìì) moderate smokers, if smoking up to 10 cigarettes/day; iii) heavy smokers if smoking more than 10 cigarettes/day.

Patients were recruited and treated in one private practice in Tirana, Albania by two operators: Marco Tallarico who performed all surgical interventions and Erta Xhanari who performed all prosthetic and maintenance procedures.

ELIGIBILITY:
Inclusion Criteria:

* Partially edentulous patient
* Bilateral edentulism in posterior maxillae (premolars and molars)
* 18 years or older
* Able to understand and sign an informed consent.
* At least 3 months after tooth extraction
* Vertical bone height at the implant sites between 2 to 6 mm
* Bone thickness at least 6 mm as measured on CBCT scan

Exclusion Criteria:

* general contraindications to implant surgery
* subjected to irradiation in the head and neck area
* immunosuppressed or immunocompromised
* treated or under treatment with intravenous amino-bisphosphonates
* poor oral hygiene and motivation
* untreated periodontal disease
* uncontrolled diabetes
* pregnant or lactating
* substance abusers
* psychiatric problems
* unrealistic expectations
* lack of opposite occluding dentition/prosthesis
* acute or chronic infection/inflammation
* augmentation/implant placement
* referred only for implant placement

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-11-01 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2019-04-02 (Actual)

PRIMARY OUTCOMES:
Prosthesis failure | Up to 5 years
  Planned prosthesis which could not be placed due to implant failure(s), loss of the prosthesis secondary to implant failure(s) or a prosthesis that had to be remade for any reasons.
Implant failure | Up to 5 years
  Implant mobility, removal of stable implants dictated by progressive marginal bone loss or infection, and implants fracture or any other mechanical complications rendering the implant unusable. The stability of each individual implant was measured with the removed prosthesis at abutment connection, at delivery definitive prostheses and at 1 year after loading, by tightening the implant abutment screws with a torque of 20 Ncm or by assessing the stability of individual crowns using the handles of two metallic instruments.
Complications | Up to 5 years
  Any technical and biological complications
Patient's preference (questionnaire) | Assessed 1 week and 1 month after surgery
  Answers: 1) the side treated with the crestal technique, 2) the side treated with the lateral technique, 3) none, both treatments were equally good, 4) none, both treatments were equally bad.

SECONDARY OUTCOMES:
Time (minutes) | The time in minutes of the surgical procedure, from the incision of the gingiva to the placement of the last stitch
  Time needs to perform the procedure, starting from the surgical incision to the delivery of the last suture, including the additional implants.
Marginal bone loss | 1 year after loading
  Assessed on digital periapical radiographs taken with the paralleling technique at implant placement, prosthesis delivery and 1 year after loading using a digital apparatus (CS 2100, Carestream Dental, Rochester, NY, US). In the case of a not properly readable radiograph, the radiograph was to be taken again. Radiographs were stored in a TIFF format with a 600 dpi resolution, in a personal computer. Peri-implant marginal bone levels were measured using the DFW 2.8 software for windows (Soredex, Tuusula, Finland). The software was calibrated for every single image using the known implant diameter. The distance between marginal bone level and implant/abutment junction, was measured at both mesial and distal sides to the nearest 0.01 mm and averaged. Bone level changes at single implants was averaged at sinus level and then at group level. Reference points for the linear measurements were: the coronal margin of the implant collar and the most coronal point of bone-to-implant contact.

CONTACTS AND LOCATIONS:
Locations (1):
- Aldent University, Tirana, Albania

IPD SHARING:
Plan to Share IPD: Undecided